CLINICAL TRIAL: NCT04817189
Title: MyRisk: Efficacy and Safety Evaluation of Oral Akynzeo® in Patients Receiving MEC at High Risk of Developing CINV Based on a Prediction Tool: A Multinational and Multicenter Study
Brief Title: Oral Akynzeo® vs Standard of Care in Preventing CINV in High-risk MEC Patients (MyRisk)
Acronym: CINV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IBA1160
Record Dates: First submitted 2021-03-01; First posted 2021-03-26 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-08

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — netupitant, palosentron drug combination; Granisetron; Palonosetron; Ondansetron; dolasetron; Tropisetron; Dexamethasone; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: interventional, open label, randomized, active controlled, parallel arms, multicenter and multinational study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg (Experimental): Oral netupitant/palonosetron (300 mg/0.50 mg) fixed-dose combination on Day 1 of each cycle.
  Dexamethasone (8 mg) will be administered on Day 1 of each cycle.
  Interventions: Drug: NEPA (300mg netupitant/0.5mg palonosetron); Drug: Dexamethasone, 8 mg (oral) or equivalent IV dose
- Standard of care + Dexamethasone 8 mg (Active Comparator): Dexamethasone (or equivalent corticosteroids) 8 mg administered by the oral route (or equivalent IV dose) on Day 1, approximately 1 hour before chemotherapy and one of the 5-HT3-RAs recommended by European Society for Medical Oncology (ESMO) and Multinational Association of Supportive Care in Cancer (MASCC) guidelines (standard of care), i.e. either:
  Granisetron, 2 mg (oral) or 1 mg (IV) OR Palonosetron, 0.5 mg (oral), 0.25mg (IV) OR Ondansetron, 16 mg (oral) or 8 mg (IV) OR Dolasetron 100 mg (oral) OR Tropisetron 5 mg (oral or IV)
  Interventions: Drug: Granisetron, 2 mg (oral) or 1 mg (IV) OR Palonosetron, 0.5 mg (oral), 0.25mg (IV) OR Ondansetron, 16 mg (oral) or 8 mg (IV) OR Dolasetron 100 mg (oral) OR Tropisetron 5 mg (oral or IV); Drug: Dexamethasone, 8 mg (oral) or equivalent IV dose

INTERVENTIONS:
Drug: NEPA (300mg netupitant/0.5mg palonosetron) — Oral netupitant/palonosetron (300 mg/0.50 mg) fixed-dose combination on Day 1 of each cycle.
  Other Names: Akynzeo® capsules
  Arms: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg
Drug: Granisetron, 2 mg (oral) or 1 mg (IV) OR Palonosetron, 0.5 mg (oral), 0.25mg (IV) OR Ondansetron, 16 mg (oral) or 8 mg (IV) OR Dolasetron 100 mg (oral) OR Tropisetron 5 mg (oral or IV) — Standard of care will be administered on Day 1 of each cycle.
  Other Names: 5-HT3 RA
  Arms: Standard of care + Dexamethasone 8 mg
Drug: Dexamethasone, 8 mg (oral) or equivalent IV dose — Dexamethasone (8 mg) will be administered on Day 1 of each cycle.
  Other Names: corticosteroid

SUMMARY:
MyRisk: Efficacy and safety evaluation of oral Akynzeo® in patients receiving MEC at high risk of developing CINV based on a prediction tool. A multinational and multicenter study.

Antiemetic guidelines recommendations are based on the emetogenic potential of the chemotherapy. Chemotherapy (CT) agents are divided in Highly, Moderately, Low and Minimally Emetogenic potential.

In addition to type of chemotherapy, several patient-related risk factors can increase the risk of CINV (chemotherapy-induced nausea and vomiting). Currently, there is limited consensus surrounding the most relevant patient risk factors that may predict the risk of CINV. Based on a recent study by Dranitsaris et al. (Dranitsaris et al. Ann Oncol. 2017 Jun 1; 28(6):1260-1267.), eight (8) predictive factors have been identified and an algorithm has been developed to incorporate these factors into the optimal selection of prophylactic antiemetics:

1. nausea and/or vomiting in the prior cycle of chemotherapy
2. use of non-prescribed antiemetics at home in the prior cycle of chemotherapy
3. platinum or anthracycline-based chemotherapy
4. age < 60 years
5. expectations for (anticipating) nausea and/or vomiting
6. <7 h of sleep the night before chemotherapy
7. history of morning sickness during previous pregnancy
8. cycle of chemotherapy (A negative association between risk and number of cycles was identified where the hazard for CINV was highest in cycles 1 and 2, with a gradual decline and plateau from cycle 3 onward).

The clinical application of this prediction tool has the potential to be an important resource for clinicians and may help to enhance patient care by optimizing the use of the antiemetics in a proactive manner.

DETAILED DESCRIPTION:
Antiemetic guideline recommendations are based on the emetogenic potential of chemotherapy and involve 4 levels of classification of intravenous chemotherapy agents, i.e., high, moderate, low and minimal; these have been accepted by major organisations. Moderate emetogenic chemotherapy (MEC) results in acute vomiting in 30% to 90% of cancer patients in the absence of antiemetic therapy. In addition to the chemotherapy type, several patient-related risk factors and clinical characteristics can increase CINV risk. These can include use of antiemetics inconsistent with international guidelines, younger age, prechemotherapy nausea, no complete CINV response in an earlier cycle, history of nausea/vomiting, (trait) anxiety, fatigue experience, and expectations of nausea/vomiting. Other studies have largely confirmed some of the key risk factors for CINV (history of vomiting during pregnancy, history of motion sickness, age, gender) and added other factors such as (chronic) alcohol consumption, body surface area, fewer hours slept the night prior to infusion, or advanced stage cancer. Currently, there is a limited consensus surrounding the most relevant patient risk factors that may predict CINV risk. Based on a recent study by Dranitsaris et al. eight predictive factors have been identified, and an algorithm has been developed to combine these patient-related risk factors into the optimal treatment of prophylactic antiemetics. These include:

1. nausea and/or vomiting in the prior cycle of chemotherapy
2. use of non-prescribed antiemetics at home in the prior cycle of chemotherapy
3. platinum or anthracycline-based chemotherapy
4. age < 60 years
5. expectations for (anticipating) nausea and/or vomiting
6. <7 h of sleep the night before chemotherapy
7. history of morning sickness during previous pregnancy
8. cycle of chemotherapy (A negative association between risk and number of cycles was identified where the hazard for CINV was highest in cycles 1 and 2, with a gradual decline and plateau from cycle 3 onward).

Akynzeo®, an oral combination of the neurokinin 1 receptor antagonists (NK1 RA), netupitant and the 5-hydroxytryptamine (HT3) receptor antagonists (5-HT3 RA), palonosetron, is recommended by guidelines for the prevention of CINV. Akynzeo® has been evaluated in a multicentre, randomised, double-blind, double-dummy phase II clinical trial at various dose ranges among 694 cisplatin-treated cancer patients from 44 sites (two countries); each NEPA (netupitant-palonosetron) dose significantly improves CINV prevention in cancer patients. Similar results were obtained in another international, randomised, double-blind and parallel group phase III clinical trial; NEPA prevented CINV in patients receiving MEC.

The current study primarily aimed to evaluate whether Akynzeo® leads to a higher response rate compared with standard care in MEC regimen-treated patients who are identified to be at high risk based on the algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years
* Patients with a risk score of ≥ 13 as calculated by the algorithm - see 3.6.3.1. Baseline/screening: VISIT 0
* Signed Informed consent
* Both sexes
* Patients with diagnosis of any cancer scheduled and intended to be treated for three consecutive cycles with a single dose of any IV MEC regimen, per cycle, including adjuvant or neo-adjuvant chemotherapy
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Use of Standard of Care defined as a 5-HT3 RA + Dexamethasone (or equivalent corticosteroid) based-regimen on day 1 of chemotherapy for CINV prevention
* Naïve and non- naïve to chemotherapy
* The enrolled women should be a) of non-childbearing potential or b) of childbearing potential using reliable contraceptive measures and having a negative urine pregnancy test done by health care team within 1-24 hours before dosing the antiemetic treatment in both arms and outcome recorded in the medical records
* Able to comply with study requirements

Exclusion Criteria:

* Patients receiving highly emetogenic chemotherapy (including anthracycline+cyclophosphamide-based chemotherapy)
* Patients receiving oral moderately emetogenic chemotherapy drugs
* Patients receiving opioids within 2 weeks prior to trial enrollment (longer use allowed)
* Use of olanzapine as prophylaxis of CINV
* Patients scheduled to receive radiotherapy concurrently with chemotherapy
* Any illness or condition that, in the opinion of the physician, may confound the results of the study or pose unwarranted risks in administering the investigational product to the patient.
* Patients with mechanical risk factors for nausea (i.e. intestinal obstruction)
* Patients with liver disease (as nausea is a common presenting symptom)
* Patients with metabolic risk factors for nausea (i.e. electrolyte imbalances causing nausea/vomiting)
* Chronic treatment with steroids (with the exception of inhaled or topical steroids)
* Pregnancy and/or breast-feeding women
* Women of childbearing potential refusing to use effective contraception during the whole study treatment and up to one month after study treatment with Akynzeo®
* Use of Standard of Care including an NK-1 RA-based regimen to prevent CINV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Molasiotis, prof., Study Chair — University of Derby
Locations (19):
- China (3):
  - Shanghai Chest Hospital, Shanghai
  - Shanghai Ninth People´s Hospital, Shanghai
  - Shanghai Obstetrics and Gynecology Hospital, Shanghai
- Czechia (2):
  - Thomayerova nemocnice, Prague
  - General University Hospital in Prague, Prague
- Germany (5):
  - Evang. Kliniken Essen-Mitte, Essen
  - Universitätsmedizin Mannheim, Mannheim
  - München Klinik Neuperlach, München
  - Frauenklinik St. Louise, Paderborn
  - Klinikum Ernst von Bergmann gemeinnützige GmbH, Potsdam
- Greece (2):
  - Sotiria General Hospital, 3rd Deúpartment of Medicine, School of Medicine, National and Kapodistrian University of Athens, Athens
  - General University Hospital of Heraklion, Heraklion
- Spain (4):
  - Complejo Hospitalario Universitario de A Coruña, A Coruña
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario de Salamanca, Salamanca
- Switzerland (2):
  - University Hospital Basel, Basel
  - Swiss Medical Network - Clinique de Genolier, Genolier
- The Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Full Analysis Set (FAS) consists of 401 (NEPA: 196, SoC: 205) randomised patients to whom study drug was dispensed. It was the primary basis for the analyses of efficacy.
Period: Overall Study
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Started | 206 | 208
Full Analysis Set (FAS) population | 196 | 205
Completed | 154 | 163
Not Completed | 52 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NEPA (300mg Netupitant/0.5mg Palonosetron) + Dexamethasone 8 mg | Standard of Care + Dexamethasone 8 mg | Total
Number analyzed (Participants) | 196 | 205 | 401
Age, Continuous [Mean (Standard Deviation); unit: year] | 62.7 (11.8) | 62.7 (11.3) | 62.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 87 | 180
  Male | 103 | 118 | 221
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
weight [Mean (Standard Deviation); unit: kg] | 73.28 (16.001) | 74.78 (17.285) | 74.05 (16.666)

OUTCOME MEASURES:

1. Primary Outcome: The Probability of Complete Responses Over Three Cycles of Chemotherapy After the Start of the MEC Administration
Description: To evaluate if the use of NEPA (netupitant and palonosetron) in patients treated with IV moderately emetogenic chemotherapy and at high risk of CINV is more effective in preventing CINV than a standard of care antiemetics over three cycles of chemotherapy.
  The primary endpoint is the probability of complete responses (no emetic episode and no rescue medication), during the overall phase (0-120h), after the start of the MEC administration over three cycles of chemotherapy. This endpoint is evaluated in patients with at least one reported cycle assessment.
  The model-based statistics of generalized linear model were used to calculate the difference in the probability to experience a "per cycle" CINV Indicators between the treatment arms.
Time Frame: At the end of all three chemotherapy cycles. The length of a cycle depends on the treatment being given (cycles range from 2 to 6 weeks).
Population: The Full Analysis Set (FAS) consists of 401 (NEPA: 196, SoC: 205) randomised patients to whom study drug was dispensed. It was the primary basis for the analyses of efficacy. Following the intent-to-treat principle, patients in the FAS population will be analysed according to the treatment to which they were randomised. The primary endpoint within the FAS was analysed based on data from 388 (NEPA: 189, SoC: 199) patients.
Measure: Number; unit: Probability of complete response
Groups:
- NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg: Oral netupitant/palonosetron (300 mg/0.50 mg) fixed-dose combination on Day 1 of each cycle.
  Dexamethasone (8 mg) will be administered on Day 1 of each cycle.
  NEPA (300mg netupitant/0.5mg palonosetron): Oral netupitant/palonosetron (300 mg/0.50 mg) fixed-dose combination on Day 1 of each cycle.
  Dexamethasone, 8 mg (oral) or equivalent IV dose: Dexamethasone (8 mg) will be administered on Day 1 of each cycle.
- Standard of care + Dexamethasone 8 mg: Dexamethasone (or equivalent corticosteroids) 8 mg administered by the oral route (or equivalent IV dose) on Day 1, approximately 1 hour before chemotherapy and one of the 5-HT3-RAs recommended by European Society for Medical Oncology (ESMO) and Multinational Association of Supportive Care in Cancer (MASCC) guidelines (standard of care), i.e. either:
  Granisetron, 2 mg (oral) or 1 mg (IV) OR Palonosetron, 0.5 mg (oral), 0.25mg (IV) OR Ondansetron, 16 mg (oral) or 8 mg (IV) OR Dolasetron 100 mg (oral) OR Tropisetron 5 mg (oral or IV)
  Granisetron, 2 mg (oral) or 1 mg (IV) OR Palonosetron, 0.5 mg (oral), 0.25mg (IV) OR Ondansetron, 16 mg (oral) or 8 mg (IV) OR Dolasetron 100 mg (oral) OR Tropisetron 5 mg (oral or IV): Standard of care will be administered on Day 1 of each cycle.
  Dexamethasone, 8 mg (oral) or equivalent IV dose: Dexamethasone (8 mg) will be administered on Day 1 of each cycle.
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 189 | 199
Probability of complete response | 0.810 | 0.718
Statistical Analysis 1: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; Test type: Superiority; p < 0.05, generalized linear model; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.12 to 2.49]; The model-based statistics were used to calculate the difference in the probability to experience a "per cycle" complete response between the treatment arms

2. Secondary Outcome: Evaluation of the Probability of Acute (0 to 24 Hours), Delayed (>24 to 120 Hours), and Overall (0-120 Hours) CINV Indicators in Each Cycle of Chemotherapy
Description: Probability of:
  * No emetic episode during the acute, delayed, and overall phase and daily in each cycle
  * No rescue medication during the acute, delayed, and overall phase and daily in each cycle
  * No significant nausea (maximum MAT scale = 2) during the acute, delayed, and overall phase and daily in each cycle;
  * No nausea (MAT scale = 0) during the acute, delayed, and overall phase and daily in each cycle;
  * Complete protection (no emetic episode, no rescue medication, and no significant nausea) during the acute, delayed, and overall phase and daily in each cycle
  Time 0 is defined as the start time of the chemotherapy administration on Day 1 of each of the three cycles.
  The model-based statistics of generalized linear model were used to calculate the difference in the probability to experience a "per cycle" CINV Indicators between the treatment arms.
Time Frame: At the end of each cycle and after all 3 chemotherapy cycles. The length of a cycle depends on the treatment being given (cycles range from 2 to 6 weeks).
Population: The model-based statistics of generalized linear model were used to calculate the difference in the probability to experience a "per cycle" CINV Indicators between the treatment arms. The probability for the Standard of Care arm is reported as the crude probability in generic cycle. The probability for the NEPA arm was calculated as the derived probability based on model odds ratio, with the model including relevant covariates.
Measure: Number; unit: Probability
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 189 | 199
Probability
  No emetic episode - acute phase | 0.983 | 0.951
  No emetic episode - delayed phase | 0.966 | 0.881
  No emetic - Day 2 | 0.981 | 0.938
  No emetic - Day 3 | 0.968 | 0.927
  No emetic - Day 4 | 0.977 | 0.938
  No emetic - Day 5 | 0.981 | 0.963
  No emetic - overall phase | 0.954 | 0.867
  No rescue medication - acute phase | 0.896 | 0.897
  No rescue medication - delayed phase | 0.848 | 0.785
  No rescue medication - Day 2 | 0.893 | 0.880
  No rescue medication - Day 3 | 0.905 | 0.872
  No rescue medication - Day 4 | 0.905 | 0.877
  No rescue medication - Day 5 | 0.910 | 0.915
  No rescue medication - overall phase | 0.824 | 0.765
  No significant nausea - acute phase | 0.868 | 0.856
  No significant nausea - delayed phase | 0.815 | 0.755
  No significant nausea - Day 2 | 0.872 | 0.817
  No significant nausea - Day 3 | 0.848 | 0.790
  No significant nausea - Day 4 | 0.847 | 0.803
  No significant nausea - Day 5 | 0.865 | 0.832
  No significant nausea - overall phase | 0.775 | 0.727
  No nausea - acute phase | 0.777 | 0.744
  No nausea - delayed phase | 0.677 | 0.576
  No nausea - Day 2 | 0.779 | 0.682
  No nausea - Day 3 | 0.749 | 0.655
  No nausea - Day 4 | 0.746 | 0.652
  No nausea - Day 5 | 0.797 | 0.703
  No nausea - overall phase | 0.637 | 0.549
  Complete protection - acute phase | 0.832 | 0.798
  Complete protection - delayed phase | 0.755 | 0.653
  Complete protection - Day 2 | 0.822 | 0.765
  Complete protection - Day 3 | 0.816 | 0.740
  Complete protection - Day 4 | 0.821 | 0.762
  Complete protection - Day 5 | 0.834 | 0.802
  Complete protection - overall phase | 0.718 | 0.624

3. Secondary Outcome: Evaluation of the Predictive Role of Potential Risk Factors in the Development of CINV Over Three Cycles of Chemotherapy
Description: Analysis of the development of CINV as a dependent variable will be performed to identify additional potential risk factors of CINV thought to be increasing the risk of CINV in patients receiving MEC.
  The outcome measure is the development of CINV, defined as any occurrence of nausea or a vomiting episode.
  The data on the development of CINV will be taken from data collection tools, patients' diaries and MASCC Antiemesis Tool (MAT).
Time Frame: as for outcome 2
Population: The Full Analysis Set (FAS). Evaluation of the predictive role of potential risk factors within the FAS was analysed based on available data from 388 (NEPA: 189, SoC: 199) patients.
  The number of patients included in the FAS population for each cycle depends on the availability of data on potential risk factors and the occurrence of nausea and/or vomiting. As the LOCF imputation method was applied for secondary endpoints, the number of participants analyzed in Cycle 1 remains lower.
Measure: Count of Participants; unit: Participants
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 189 | 199
Participants
  Cycle 1 - Any occurrence of nausea or a vomiting episode: number analyzed (Participants) | 188 | 198
  Cycle 1 - Any occurrence of nausea or a vomiting episode | 77 | 97
  Cycle 2 - Any occurrence of nausea or a vomiting episode | 71 | 90
  Cycle 3 - Any occurrence of nausea or a vomiting episode | 65 | 86
Statistical Analysis 1: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; The hypothesis states that the potential risk factor of < 7 h of sleep the night before chemotherapy increases the risk of CINV, defined as any occurrence of nausea or a vomiting episode. This potential risk factor was included in the generalized linear model as covariate, and its effect was evaluated using odds ratios; Test type: Superiority; p = 0.412, generalized linear model; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.68 to 1.17] — Reference category is set to Sleep ≥ 7 h, compared to Sleep < 7 h
Statistical Analysis 2: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; The hypothesis states that the potential risk factor of History of any nausea and vomiting such as motion sickness, vestibular dysfunction, … increases the risk of CINV, defined as any occurrence of nausea or a vomiting episode. This potential risk factor was included in the generalized linear model as covariate, and its effect was evaluated using odds ratios; Test type: Superiority; p = 0.592, generalized linear model; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.71 to 1.80] — Reference category is set to Without history, compared to With history
Statistical Analysis 3: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; The hypothesis states that the potential risk factor of Anticipatory nausea and/or vomiting increases the risk of CINV, defined as any occurrence of nausea or a vomiting episode. This potential risk factor was included in the generalized linear model as covariate, and its effect was evaluated using odds ratios; Test type: Superiority; p = 0.458, generalized linear model; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.80 to 1.65] — Reference category is set to No anticipatory, compared to Anticipatory
Statistical Analysis 4: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; The hypothesis states that the potential risk factor of Anxiety over the past 24hrs increases the risk of CINV, defined as any occurrence of nausea or a vomiting episode. This potential risk factor was included in the generalized linear model as covariate, and its effect was evaluated using odds ratios; Test type: Superiority; p = 0.663, generalized linear model; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.75 to 1.56] — Reference category is set to No anxiety, compared to Anxiety
Statistical Analysis 5: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; The hypothesis states that the potential risk factor of Alcohol intake (>= 10 units per week vs < 10 units per week) increases the risk of CINV, defined as any occurrence of nausea or a vomiting episode. This potential risk factor was included in the generalized linear model as covariate, and its effect was evaluated using odds ratio; Test type: Superiority; p = 0.691, generalized linear model; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.46 to 1.68] — Reference category is set to < 10 units per week, compared to >= 10 units per week
Statistical Analysis 6: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; The hypothesis states that the potential risk factor of Gender increases the risk of CINV, defined as any occurrence of nausea or a vomiting episode. This potential risk factor was included in the generalized linear model as covariate, and its effect was evaluated using odds ratios; Test type: Superiority; p = 0.037, generalized linear model; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.02 to 2.14] — Reference category is set to Male, compared to Female
Statistical Analysis 7: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; The hypothesis states that the potential risk factor of Fatigue experience (symptom) increases the risk of CINV, defined as any occurrence of nausea or a vomiting episode. This potential risk factor was included in the generalized linear model as covariate, and its effect was evaluated using odds ratios; Test type: Superiority; p = 0.514, generalized linear model; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.84 to 1.42] — Reference category is set to No fatigue experience, compared to Fatigue experience
Statistical Analysis 8: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; The hypothesis states that the potential risk factor of Smoking status increases the risk of CINV, defined as any occurrence of nausea or a vomiting episode. This potential risk factor was included in the generalized linear model as covariate, and its effect was evaluated using odds ratios; Test type: Superiority; p = 0.127, generalized linear model; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.52 to 1.08] — Reference category is set to Non smoker, compared to Former smoker or smoker
Statistical Analysis 9: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; The hypothesis states that the potential risk factor of Weight increases the risk of CINV, defined as any occurrence of nausea or a vomiting episode. This potential risk factor was included in the generalized linear model as covariate, and its effect was evaluated using odds ratios; Test type: Superiority; p = 0.014, generalized linear model; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.77 to 0.97] — The OR was calculated as the change in weight per 10 kg

4. Secondary Outcome: Evaluation of the Safety Profile of the Antiemetic Drug Over Three Cycles of Chemotherapy - the Frequency of Adverse Events (AE)
Description: An overall summary of adverse events (AE) will be presented, including the frequency of patients with:
  * Any treatment-emergent adverse event
  * Any treatment-emergent adverse event related to a study drug
  * Any treatment-emergent adverse event leading to chemotherapy dose reductions or interruptions
  * Any treatment-emergent serious adverse event
  All AEs will be summarized by their:
  * Severity
  * Seriousness
  * Relationship to a drug
Time Frame: At the end of all 3 chemotherapy cycles. The length of a cycle depends on the treatment being given (cycles range from 2 to 6 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
Participants
  Patients with any TEAE | 150 | 150
  Patients with any TEAE related to a study drug | 37 | 38
  Patients with any TEAE leading to chemotherapy dose reductions | 6 | 11
  Patients with any TEAE leading to treatment discontinuation | 5 | 7
  Patients with any serious TEAE | 22 | 23
  Patients with any severe TEAE | 26 | 32
  Patients with on treatment death due to TEAE | 2 | 2

5. Secondary Outcome: Evaluation of the Safety Profile of the Antiemetic Drug Over Three Cycles of Chemotherapy - Percentage of Participants With Adverse Events
Description: An overall summary of adverse events (AE) will be presented, including the percentage of patients with:
  * Any treatment-emergent adverse event
  * Any treatment-emergent adverse event related to a study drug
  * Any treatment-emergent adverse event leading to chemotherapy dose reductions or interruptions
  * Any treatment-emergent serious adverse event
  All AEs will be summarized by their:
  * Severity
  * Seriousness
  * Relationship to a drug
Time Frame: as for outcome 4
Measure: Number; unit: percentage of patients
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
percentage of patients
  Patients with any TEAE | 76.5 | 73.2
  Patients with any TEAE related to a study drug | 18.9 | 18.5
  Patients with any TEAE leading to chemotherapy dose reductions | 3.1 | 5.4
  Patients with any TEAE leading to treatment discontinuation | 2.6 | 3.4
  Patients with any serious TEAE | 11.2 | 11.2
  Patients with any severe TEAE | 13.3 | 15.6
  Patients with on treatment death due to TEAE | 1.0 | 1.0

6. Secondary Outcome: Number of Participants With Discontinuations Due to Adverse Events
Description: The frequency of discontinuations due to adverse events (AE) will be presented.
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
Participants | 5 | 7

7. Secondary Outcome: Percentage of Participants With Discontinuations Due to Adverse Events
Description: The percentage of patients with discontinuations due to adverse events (AE) will be presented.
Time Frame: as for outcome 4
Measure: Number; unit: percentage of patients
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
percentage of patients | 2.6 | 3.4

8. Secondary Outcome: Number of Participants With Death Due to Adverse Events
Description: The frequency of on treatment deaths due to adverse events (AE) will be presented.
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
Participants | 2 | 2

9. Secondary Outcome: Percentage of Participants With Death Due to Adverse Events
Description: The percentage of patients with on treatment death due to adverse events (AE) will be presented.
  All AEs leading to on treatment death will be summarized by their:
  * Severity
  * Seriousness
  * Relationship to a drug
Time Frame: as for outcome 4
Measure: Number; unit: percentage of patients
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
percentage of patients | 1.0 | 1.0

10. Secondary Outcome: Exploration of the Effect of CINV on Daily Activities and Quality of Life in Patients Receiving Moderately-emetogenic Chemotherapy Over Three Cycles of Chemotherapy
Description: Evaluation of the effect of CINV on daily activities and quality of life that will be measured by using the Functional Living Index-Emesis (FLIE) questionnaire, a validated, nausea and vomiting specific, patient-reported outcome instrument.
  The Functional Living Index-Emesis (FLIE) has 18 questions. These questions are divided into two domains: Nausea (questions 1-9) and Vomiting (questions 10-18).
  The minimum score for any question is 0 and the maximum score is 100. Higher scores indicate less impairment on daily life as a result of nausea or vomiting.
  The model-based statistics of generalized linear model were used to calculate the difference in the score "per cycle" between the treatment arms.
Time Frame: At the end of chemotherapy cycles. The length of a cycle depends on the treatment being given (cycles range from 2 to 6 weeks).
Population: Full analysis set. Patients with evaluable data in cycle 1 and eligible for imputation, using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: FLIE score
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 189 | 199
FLIE score
  After cycle 1 - FLIE score | 115.14 (17.152) | 111.10 (21.134)
  After cycle 2 - FLIE score | 115.78 (18.022) | 112.10 (19.919)
  After cycle 3 - FLIE score | 114.74 (19.356) | 111.24 (21.772)
Statistical Analysis 1: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; Test type: Superiority; p < 0.05, generalized linear model; Mean Difference (Net) = 3.5, 95% CI 2-sided [0.05 to 6.96]; The model-based statistics were used to calculate the difference in the score "per cycle" between the treatment arms

11. Secondary Outcome: Evaluation of Resource Utilization and Health Economic Outcome - Number of Days With Rescue Medication Administered for the Treatment of CINV
Description: Health economic endpoint, the number of days with rescue medication administered for the treatment of CINV, will be evaluated during the study cycles
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
Number of days
  cycle 1 | 0.5 (1.20) | 0.5 (1.13)
  Cycle 2 | 0.4 (1.20) | 0.6 (1.26)
  Cycle 3 | 0.5 (1.28) | 0.5 (1.22)

12. Secondary Outcome: Evaluation of Resource Utilization and Health Economic Outcome - Daily Doses of Rescue Medication Administered for the Treatment of CINV
Description: Health economic endpoint, the daily doses of rescue medication administered for the treatment of CINV, will be evaluated during the study cycles
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: Doses of medication per cycle
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
Doses of medication per cycle
  Cycle 1 | 16.3 (68.53) | 46.3 (343.13)
  Cycle 2 | 13.7 (57.0) | 19.9 (70.87)
  Cycle 3 | 24.7 (99.48) | 17.5 (74.24)

13. Secondary Outcome: Evaluation of Resource Utilization and Health Economic Outcome - the Number of Re-hydration Bags
Description: Health economic endpoint, the number of re-hydration bags given for at least grade 2 vomiting (more details below), will be evaluated during the study cycles
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of bags
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
Number of bags
  Cycle 1 | 0 (0.00) | 0 (0.20)
  Cycle 2 | 0 (0.00) | 0 (0.15)
  Cycle 3 | 0 (0.00) | 0 (0.00)

14. Secondary Outcome: Evaluation of Resource Utilization and Health Economic Outcome - the Number of Days of Unplanned Hospitalisations
Description: Health economic endpoint, the number of days of unplanned hospitalizations related to CINV, will be evaluated during the study cycles
  All hospitalizations will be summarized according to the department of hospitalization (type of ward)
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: days of hospitalization
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
days of hospitalization
  Cycle 1 | 0 (0.07) | 0.1 (0.75)
  Cycle 2 | 0 (0.23) | 0 (0.30)
  Cycle 3 | 0 (0.00) | 0 (0.38)

15. Secondary Outcome: Evaluation of Resource Utilization and Health Economic Outcome - the Number of Outpatient Physician Visits
Description: Health economic endpoint, the number of outpatient physician visits and health care consultations due to CINV (e.g., general practitioner), will be evaluated during the study cycles
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of outpatient visits
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
Number of outpatient visits
  Cycle 1 | 0 (0.07) | 0 (0.16)
  Cycle 2 | 0 (0.08) | 0 (0.15)
  Cycle 3 | 0 (0.00) | 0 (0.00)

16. Secondary Outcome: Evaluation of Resource Utilization and Health Economic Outcome - the Number of Unplanned Laboratory Test
Description: Health economic endpoint, the number of unplanned laboratory test including those at unplanned hospitalizations due to CINV, will be evaluated during the study cycles
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of unplanned tests
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
Number of unplanned tests
  Cycle 1 | 0 (0.07) | 0.1 (0.46)
  Cycle 2 | 0 (0.15) | 0 (0.16)
  Cycle 3 | 0 (0.00) | 0 (0.23)

17. Secondary Outcome: Evaluation of Resource Utilization and Health Economic Outcome - Discontinuation of Chemotherapy Treatment Due to CINV
Description: Health economic endpoint, the number of discontinuations of chemotherapy treatment due to CINV, will be evaluated during the study cycles
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
Participants
  Cycle 1 | 1 | 0
  Cycle 2 | 1 | 1
  Cycle 3 | 0 | 0

18. Secondary Outcome: Evaluation of Resource Utilization and Health Economic Outcome - the Number of Delays of Chemotherapy Administration Due to CINV
Description: Health economic endpoint, the number of delays of chemotherapy administration due to CINV, will be evaluated during the study cycles.
  Delays will be observed after the first administration of Cycle 1 for Cycles 2 and 3.
Time Frame: At the start of cycles 2 and 3. The length of a cycle depends on the treatment being given (cycles range from 2 to 6 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
Participants
  Cycle 2 | 0 | 2
  Cycle 3 | 0 | 3

19. Secondary Outcome: Evaluation of Resource Utilization and Health Economic Outcome - the Average Length of Delay of Chemotherapy Administration Due to CINV
Description: Health economic endpoint, the average length of delay (in days) of chemotherapy administration due to CINV, will be evaluated during the study cycles.
  Delays will be observed after the first administration of Cycle 1 for Cycles 2 and 3.
Time Frame: as for outcome 18
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
Days
  Cycle 2 | 0 (0) | 7 (0.00)
  Cycle 3 | 0 (0) | 7.7 (1.15)

20. Secondary Outcome: Evaluation of Resource Utilization and Health Economic Outcome - Days of Absence From Work
Description: Health economic endpoint, the number of days of absence from work, will be evaluated during the study cycles
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 196 | 205
Days
  Cycle 1 | 3 (3.08) | 5.7 (4.16)
  Cycle 2 | 1 (0.00) | 4.3 (3.59)
  Cycle 3 | 2.4 (1.34) | 7.0 (2.83)

21. Secondary Outcome: Evaluation of Acute (0 to 24 Hours), Delayed (>24 to 120 Hours), and Overall (0-120 Hours) CINV Indicators in Each Cycle of Chemotherapy
Description: Number of vomiting episodes during the acute, delayed, and overall phase in each cycle
  Time 0 is defined as the start time of the chemotherapy administration on Day 1 of each of the three cycles.
  The model-based statistics of generalized linear model were used to calculate the difference in the number of vomiting episodes "per cycle" between the treatment arms.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Number of vomiting episodes
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
Number analyzed (Participants) | 189 | 199
Number of vomiting episodes
  Cycle 1 acute phase - Number of vomiting episodes | 0.04 (0.300) | 0.09 (0.494)
  Cycle 2 acute phase - Number of vomiting episodes | 0.04 (0.316) | 0.10 (0.508)
  Cycle 3 acute phase - Number of vomiting episodes | 0.05 (0.422) | 0.11 (0.601)
  Cycle 1 delayed phase - Number of vomiting episodes | 0.08 (0.425) | 0.46 (1.579)
  Cycle 2 delayed phase - Number of vomiting episodes | 0.06 (0.440) | 0.35 (1.424)
  Cycle 3 delayed phase - Number of vomiting episodes | 0.10 (0.701) | 0.36 (1.507)
  Cycle 1 day 2 - Number of vomiting episodes | 0.03 (0.230) | 0.19 (0.893)
  Cycle 2 day 2 - Number of vomiting episodes | 0.02 (0.177) | 0.10 (0.481)
  Cycle 3 day 2 - Number of vomiting episodes | 0.05 (0.422) | 0.18 (0.969)
  Cycle 1 day 3 - Number of vomiting episodes | 0.07 (0.433) | 0.20 (0.825)
  Cycle 2 day 3 - Number of vomiting episodes | 0.09 (0.690) | 0.11 (0.579)
  Cycle 3 day 3 - Number of vomiting episodes | 0.09 (0.543) | 0.17 (0.777)
  Cycle 1 day 4 - Number of vomiting episodes | 0.05 (0.449) | 0.14 (0.593)
  Cycle 2 day 4 - Number of vomiting episodes | 0.10 (0.670) | 0.11 (0.556)
  Cycle 3 day 4 - Number of vomiting episodes | 0.10 (0.594) | 0.17 (0.769)
  Cycle 1 day 5 - Number of vomiting episodes | 0.05 (0.431) | 0.07 (0.438)
  Cycle 2 day 5 - Number of vomiting episodes | 0.06 (0.480) | 0.10 (0.527)
  Cycle 3 day 5 - Number of vomiting episodes | 0.07 (0.506) | 0.15 (0.792)
  Cycle 1 overall phase - Number of vomiting episodes | 0.11 (0.516) | 0.55 (1.804)
  Cycle 2 overall phase - Number of vomiting episodes | 0.10 (0.585) | 0.45 (1.760)
  Cycle 3 overall phase - Number of vomiting episodes | 0.15 (0.837) | 0.47 (1.909)
Statistical Analysis 1: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; Test type: Superiority; p < 0.05, generalized linear model; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.13 to 0.01] — Number of vomiting episodes - acute phase
Statistical Analysis 2: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; Test type: Superiority; p < 0.05, generalized linear model; Mean Difference (Net) = -0.31, 95% CI 2-sided [-0.50 to -0.12] — Number of vomiting episodes - delayed phase
Statistical Analysis 3: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; Test type: Superiority; p < 0.05, generalized linear model; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.21 to -0.02]; Number of vomiting episodes - Day 2
Statistical Analysis 4: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; Test type: Superiority; p < 0.05, generalized linear model; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.17 to 0.04] — Number of vomiting episodes - Day 3
Statistical Analysis 5: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; Test type: Superiority; p < 0.05, generalized linear model; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.16 to 0.05] — Number of vomiting episodes - Day 4
Statistical Analysis 6: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; Test type: Superiority; p < 0.05, generalized linear model; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.13 to 0.05] — Number of vomiting episodes - Day 5
Statistical Analysis 7: Comparison: NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg vs Standard of care + Dexamethasone 8 mg; Test type: Superiority; p < 0.05, generalized linear model; Mean Difference (Net) = -0.37, 95% CI 2-sided [-0.60 to -0.14] — Number of vomiting episodes - overall phase

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the date of informed consent to Day 5 of Cycle 3 (approximately 6.3 weeks). The longest time period was 17.6 weeks. The time differes per the days of the chemotherapy cycle.
Arm/Group | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg | Standard of care + Dexamethasone 8 mg
All-Cause Mortality (participants affected / at risk) | 2/196 | 2/205
Serious Adverse Events (participants affected / at risk) | 22/196 | 23/205
Other Adverse Events (participants affected / at risk) | 150/196 | 150/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg (N=196) | Standard of care + Dexamethasone 8 mg (N=205)
neutropenia (Blood and lymphatic system disorders) | 6 | 5
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Death (General disorders) | 2 | 2
Pyrexia (General disorders) | 3 | 1
General physical health deterioration (General disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hyper-transaminasaemia (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Abscess oral (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Ludwig angina (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Aphasia (Nervous system disorders) | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 1 | 0
Hemianopia (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Antibiotic therapy (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NEPA (300mg netupitant/0.5mg palonosetron) + Dexamethasone 8 mg (N=196) | Standard of care + Dexamethasone 8 mg (N=205)
Neutropenia (Blood and lymphatic system disorders) | 8 | 7
Anaemia (Blood and lymphatic system disorders) | 3 | 8
Leukocytosis (Blood and lymphatic system disorders) | 1 | 4
Vertigo (Ear and labyrinth disorders) | 4 | 7
Diarrhoea (Gastrointestinal disorders) | 40 | 48
Constipation (Gastrointestinal disorders) | 41 | 29
Abdominal pain (Gastrointestinal disorders) | 19 | 25
Nausea (Gastrointestinal disorders) | 15 | 17
Dyspepsia (Gastrointestinal disorders) | 9 | 6
Dry mouth (Gastrointestinal disorders) | 8 | 6
Abdominal discomfort (Gastrointestinal disorders) | 3 | 10
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2
Stomatitis (Gastrointestinal disorders) | 4 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 6
Eructation (Gastrointestinal disorders) | 5 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4
Hypoaesthesia oral (Gastrointestinal disorders) | 2 | 4
Abdominal distension Flatulence (Gastrointestinal disorders) | 4 | 1
Flatulence (Gastrointestinal disorders) | 0 | 4
Oral pain (Gastrointestinal disorders) | 0 | 4
Paraesthesia oral (Gastrointestinal disorders) | 0 | 4
Fatigue (General disorders) | 54 | 46
Asthenia (General disorders) | 25 | 21
General physical health deterioration (General disorders) | 3 | 12
Pain (General disorders) | 6 | 7
Pyrexia (General disorders) | 4 | 7
Oedema peripheral (General disorders) | 1 | 8
Chest pain (General disorders) | 2 | 4
Chills (General disorders) | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 23 | 30
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 3
Limb discomfort (Musculoskeletal and connective tissue disorders) | 6 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Paraesthesia (Nervous system disorders) | 33 | 26
Dizziness (Nervous system disorders) | 24 | 15
Neuropathy peripheral (Nervous system disorders) | 15 | 20
Headache (Nervous system disorders) | 18 | 15
Hypoaesthesia (Nervous system disorders) | 11 | 20
Neurotoxicity (Nervous system disorders) | 10 | 8
Dysgeusia (Nervous system disorders) | 8 | 7
Polyneuropathy (Nervous system disorders) | 6 | 7
Somnolence (Nervous system disorders) | 7 | 5
Cold dysaesthesia (Nervous system disorders) | 4 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 2
Taste disorder (Nervous system disorders) | 2 | 4
Insomnia (Psychiatric disorders) | 4 | 8
Restlessness (Psychiatric disorders) | 2 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 12
Erythema (Skin and subcutaneous tissue disorders) | 5 | 7
Rash (Skin and subcutaneous tissue disorders) | 9 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 5
Peripheral coldness (Vascular disorders) | 5 | 4
Hypotension (Vascular disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/89/NCT04817189/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT04817189/SAP_001.pdf